CLINICAL TRIAL: NCT05888922
Title: International Phase III, Multi Center, Randomized, Double Blind, Placebo and Active Controlled and Parallel Group Clinical Trial to Evaluate the Efficacy and Safety of Oral Minoxidil 1 mg in Female Patients With Androgenetic Alopecia
Brief Title: Evaluation of Efficacy and Safety of Oral Minoxidil 1 mg in Female Androgenetic Alopecia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Industrial Farmacéutica Cantabria, S.A. (Industry)
Collaborators: Bioskin GmbH (Industry); BioClever 2005 S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P22112a
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Androgenetic Alopecia; Female Pattern Baldness
Keywords: Androgenetic alopecia; Female Pattern Baldness; FAGA; Minoxidil
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active group (Experimental): Oral minoxidil 1 mg (1 tablet, OD) + topical vehicle solution (1 ml, BID)
  Interventions: Drug: Minoxidil Tablets; Drug: Vehicle solution
- Control group (Active Comparator): Oral placebo (1 tablet, OD) + topical 2% Minoxidil solution (1 ml, BID)
  Interventions: Drug: Minoxidil Topical; Drug: Placebo oral tablet
- Placebo group (Placebo Comparator): oral placebo (1 tablet, OD) + topical vehicle solution (1 ml, BID)
  Interventions: Drug: Placebo oral tablet; Drug: Vehicle solution

INTERVENTIONS:
Drug: Minoxidil Tablets — The clinical trial will use a block randomization scheme to assign those eligible patients to one of the three arms of the study treatment on a 2:2:1 ratio. All patients will be given a kit with oral tablets (active/placebo) 1 tablet to be taken once a day and a topical solution (active comparator/vehicle) to be applied 1 ml twice daily.
  Arms: Active group
Drug: Minoxidil Topical — The clinical trial will use a block randomization scheme to assign those eligible patients to one of the three arms of the study treatment on a 2:2:1 ratio. All patients will be given a kit with oral tablets (active/placebo) 1 tablet to be taken once a day and a topical solution (active comparator/vehicle) to be applied 1 ml twice daily.
  Arms: Control group
Drug: Placebo oral tablet — The clinical trial will use a block randomization scheme to assign those eligible patients to one of the three arms of the study treatment on a 2:2:1 ratio. All patients will be given a kit with oral tablets (active/placebo) 1 tablet to be taken once a day and a topical solution (active comparator/vehicle) to be applied 1 ml twice daily.
  Arms: Control group; Placebo group
Drug: Vehicle solution — The clinical trial will use a block randomization scheme to assign those eligible patients to one of the three arms of the study treatment on a 2:2:1 ratio. All patients will be given a kit with oral tablets (active/placebo) 1 tablet to be taken once a day and a topical solution (active comparator/vehicle) to be applied 1 ml twice daily.
  Arms: Active group; Placebo group

SUMMARY:
The goal of this clinical trial is to learn about oral minoxidil 1mg in the treatment of women with androgenetic alopecia, a type of hormone-imbalanced hair loss.

The main questions to answer are to know about that minoxidil 1mg is as effective as minoxidil 2% topical solution (comparator product) and is more effective than placebo; and to ensure treatment with oral minoxidil is safe.

Participants will be assigned randomly to receive one of the following treatment combinations:

* the test product (oral minoxidil 1 mg, once/day) and the vehicle solution (vehicle means it looks like the comparator product, but it does not contain an active ingredient, 2 times/day), or
* the placebo tablet (placebo means it looks like the test product, but it does not contain an active ingredient, once/day) and the comparator product (2% minoxidil solution, 2 times/day), or
* the placebo tablet (once/day) and the vehicle solution (2 times/day).

The clinical trial will take up to 36 weeks. During this time, patients will come to the clinical trial centre for 5 times for examinations and will be called by phone twice. At the visits, the following examinations will be performed: photos of the hair will be taken to determine hair density, assessment of changes in scalp hair growth, measurement of blood pressure, pulse, and body temperature, a physical examination, blood withdrawal to determine any abnormalities in the blood, urine sampling and analysis, performance of ECG, and evaluation of hypertrichosis (i.e., excessive hair growth over the body). Furthermore, patients will be asked daily whether they had experienced any side effects or took any new medications (or changed the dose of a known medication) or underwent any medical procedure. Also, women of childbearing potential must undergo pregnancy tests in blood and urine.

DETAILED DESCRIPTION:
This is a phase III, multi center, randomized, double blind, placebo and active controlled parallel group design clinical trial to evaluate the efficacy and safety of oral minoxidil 1 mg for the treatment of AGA in female* patients aged 18 years or older, with general good health (i.e., with no history of cardiovascular disorders, or any other clinically significant disease) and without any dermatological disorders (e.g., of the scalp in the target region at Visit 1/Screening with the possibility of interfering with the application of the IPs or examination method).

Patients must show and have a history of hair density reduction in the centroparietal area of the scalp, as classified by the Sinclair Scale (Sinclair Scale 2-4).

It is planned that approximately 520 adult female patients with FAGA from 20 trial centers across 4 countries (Germany, Spain, Italy, and Portugal) will enter the clinical trial.

Eligible patients will be randomly assigned in a ratio 2:2:1 (active: control: placebo) to one of the following 3 treatment groups:

1. Active group: oral minoxidil 1 mg (1 tablet, once daily [OD]) + topical vehicle solution (1 ml, twice daily [BID])
2. Control group: oral placebo (1 tablet, OD) + topical 2% minoxidil solution (1 ml, BID)
3. Placebo group: oral placebo (1 tablet, OD) + topical vehicle solution (1 ml, BID)

At Visit 2/Baseline, patients will receive three boxes containing 5 blister packs of 10 tablets each (a total of 50 tablets) and 4 bottles of IP solution containing 60 ml of 2% minoxidil solution each to cover 12 weeks (±7 days) of clinical trial treatment. The patients will be instructed how to apply the IPs. The first topical IP treatment will be performed under supervision at the clinical trial center, and then treatments will be performed by the patients at home (also the intake of the first tablet), as follows: Patients will administer the assigned IPs daily for 6 months-one tablet orally OD (in the evening/at night [preferably before going to bed to minimize anti hypertensive side effects]) and 2 ml assigned solution topically to the scalp BID (two topical applications of 1 ml each, to be performed at least 8 hours apart). Each patient will be requested to record date and time of treatments in an electronic patient dosing diary (hereinafter called "electronic diary [e-diary]"). At the next planned clinical trial center visit (Visit 4/Week 12), the patients will receive a new batch of clinical trial treatment for the next 12 weeks.

The clinical trial consists of a screening period (up to approximately 8 weeks, Week 8 to Day -2), a 6 month treatment period (Week 0 to 24), and a 4 week follow up period (Week 25 to 28).

It is planned to have five clinical trial center visits (Visit 1/Screening, Visit 2/Baseline, Visit 4/Week 12, Visit 6/Week 24, and Visit 7/Week 28) and two safety phone calls (Visit 3/Week 4 and Visit 5/Week 18) during the course of the clinical trial; unscheduled visits may be needed per the discretion of the investigator. Efficacy and safety will be evaluated and compared among the three treatment groups.

The duration of clinical trial participation for each patient will be approximately up to 36 weeks.

At the screening visit, the clinical trial requirements and procedures will be reviewed. Written informed consent will be obtained prior to the initiation of any clinical trial related procedures (including washout). Once informed consent has been signed, the patient will be assigned a patient number. The suitability of the patient hair color (sufficient contrast with the scalp) for re-detection of the target area will be assessed by means of the TrichoLab Virtual Tattoo®technology which includes the taking of two microphotographs.

If applicable, qualified patients can washout from prohibited medications or treatments prior to Visit 2/Baseline (after obtaining written informed consent). Patients must return to the clinical trial center after washout for completion of screening procedures.

The following screening procedures must take place up to within 8 weeks of Visit 2/Baseline:

Demographics, inclusions/exclusion criteria, relevant medical and relevant surgical history of the past 5 years, and prior as well as concomitant medications and therapies of the last 12 months will be reviewed. The patient's FAGA will be classified using the Sinclair Scale. A brief physical examination, vital signs (blood pressure, pulse rate, body temperature), height and weight, safety laboratory tests (hematology, clinical chemistry, and urinalysis), serum pregnancy test (only for women of childbearing potential [WOCBP]), and 12 lead ECG will be performed. AEs will be recorded, as applicable. Preliminary patient eligibility will be assessed, and, if applicable, the patient will be scheduled for Visit 2/Baseline.

During the clinical trial, safety will be assessed through physical examination, vital signs, weight, 12 lead ECG, and safety laboratory tests (hematology, clinical chemistry, and urinalysis) at each clinical trial center visit, except for safety laboratory which will not be performed at Visit 7/Week 28.

Hypertrichosis evaluation will be performed at Visit 2/Baseline, Visit 4/Week 12, Visit 6/Week 24 (end of treatment [EoT)/early termination visit [ETV]), and Visit 7/Week 28.

AEs, as well as concomitant medication, and procedures will be documented from the time point the patient has signed the informed consent form (ICF) until the end of clinical trial.

For all WOCBP, a urine pregnancy test will be performed at Visit 2/Baseline, Visit 4/Week 12, and Visit 6/Week 24.

During the clinical trial, efficacy will be determined based on quantitative hair measurements of Target Area non-vellus Hair Counts (TAHC), Target Area non vellus Hair Width (TAHW), and Target Area non vellus Hair Density (TAHD) at each clinical trial center visit except for Visit 1/Screening and Visit 7/Week 28. TAHC, TAHW, and TAHD will be determined by using TrichoLAB Hair-to-hair Matching® technology and digital image analysis.

In addition, hair growth assessments will be performed by the investigator at Visit 4/Week 12 and Visit 6/Week 24 (Investigator's Global Assessment [IGA, 7 point scale]), using the standardized approved global photo of the patient's scalp taken at Visit 2/Baseline. Furthermore, the patient's quality of life will be assessed by means of a patient self-questionnaire (Women's Androgenetic Alopecia Quality of Life [WAA QoL] at Visit 2/Baseline Visit 4/Week 12 and Visit 6/Week 24.

Statistical analyses will be conducted based on the available data, without using techniques for inputting missing values, but describing the number of missing values for each analysis.

All statistical tests will be performed at a significance level of α = 0.01, unless specifically stated otherwise.

Prior to the database closure, a statistical analysis plan (SAP) will be approved in which the whole strategy of data analysis will be described in detail.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 years or older, with general good health (i.e., with no history of cardiovascular disorders, or any other clinically significant disease).
2. Diagnosed with FAGA, based on a discernible decrease in hair density (Sinclair Scale 2-4) in the centroparietal area of the scalp.
3. Hair color of patient provides sufficient contrast with the scalp and as confirmed by TrichoLab Virtual Tattoo® technology at Screening/Visit 1.
4. A personally signed and dated informed consent document indicating that the patient, has been informed of all pertinent aspects of the clinical trial.
5. Negative serum pregnancy test at Visit 1/Screening and negative urine pregnancy test at Visit 2/Baseline for women of child-bearing potential (WOCBP).
6. WOCBP must either be permanently sterile1 or agree to use a highly effective birth control method (failure rate ˂1% per year when used consistently and correctly) throughout the clinical trial and for at least 2 weeks after last administration of IPs.

   Gestagens with antiandrogen properties (e.g., cyproterone acetate, dienogest) are allowed if treatment is stable since the last 6 months prior to Visit 2/Baseline and if used as contraceptive and planned to be continued throughout the clinical trial duration.
7. Patients willing to maintain the same hairstyle (color and hair regimen) throughout the clinical trial. Hair length must remain of sufficient length to not affect determination of hair density and patient should discuss with clinical trial personnel before changing from Visit 2/Baseline.
8. Patient is willing to maintain the same depilatory habits and intervals regarding facial or body hair before each visit throughout duration of the clinical trial.
9. Patient is willing and able to comply with scheduled visits, treatment plan, laboratory tests and other clinical trial procedures, including daily e diary recordings by the patient using an own electronic device (e.g., tablet, smartphone, personal computer) and an internet connection during the clinical trial.

Exclusion Criteria:

1. Known hypersensitivity or known allergy to minoxidil or to any of the other components of the products.
2. Pregnancy or pregnancy desire during the clinical trial.
3. Breastfeeding/Nursing women.
4. Any diagnosed treated or untreated hypertension (or blood pressure values >150 mmHg systolic / >95 mmHg diastolic) as determined at Visit 1/Screening, and/or history/signs of known cardiovascular diseases (including but not limited to cardiac ischemia, congestive heart failure, cardiac arrhythmia), and patients with pathologies or punctual situations that might either be caused by or increase the risk of cardiac disorders.
5. Patients with any dermatological disorders of the scalp in the target region at Visit 1/Screening with the possibility of interfering with the application of the IPs or examination method, such as

   1. Active moderate or severe seborrheic dermatitis under chronic treatment, abrasion, actinic keratosis, or inflammatory disorders, or
   2. any local infection of the skin/subcutaneous tissues of the head within the previous 3 months, or
   3. any documented history of active atopic dermatitis or psoriasis in the scalp within the previous 6 months.
   4. any other types of alopecia (e.g., alopecia areata or scarring alopecia) at any time point or diffuse telogen effluvium, trichotillomania, or other pathological hair loss conditions/diseases other than AGA in the last 3 months at the discretion of the investigator).
6. Patients who had hair transplant surgery at any time.
7. Patients who had hair weaving, or any other hair extension methods within the last 6 months prior to Visit 2/Baseline.
8. Clinically significant abnormal laboratory values or ECG findings (if applicable) at Visit 1/Screening indicative of physical illness, according to investigator assessment.
9. Both creatinine and eGFR above upper limit of normal at Visit 1/Screening.
10. Relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, or neurological diseases that in the opinion of the investigator may interfere with the aim of the clinical trial.
11. Patient has used any of the following topical preparations or procedures on the scalp:

    1. Topical scalp treatments for hair growth, including minoxidil within the last 6 months prior to Visit 2/Baseline; or hormone therapy, antiandrogens, or other agents that are known to affect hair growth within 12 weeks prior to Visit 2/Baseline.
    2. Topical scalp treatments that might have had ancillary effect on hair growth including, but not limited to, corticosteroids, pimecrolimus, and tacrolimus within the last 4 weeks prior to Visit 2/Baseline.
    3. Topical scalp over the counter (OTC) or cosmetic treatments known or reasonably believed to affect hair growth (e.g., brands such as Maxilene®, Nioxin®, Foltene®, etc.) or hair health or hair growth products with saw palmetto, copper, etc. within the last 4 weeks prior to Visit 2/Baseline.
    4. Light or laser treatment or microneedling of scalp within the last 6 months prior to Visit 2/Baseline.
    5. Platelet rich plasma (PRP) procedure on the scalp within the last 6 months prior to Visit 2/Baseline.
12. Patient has used the following systemic medications or procedures:

    1. Zidovudine, cyclosporine, diazoxide, phenytoin, systemic interferon, psoralens, streptomycin, penicillamine, benoxaprofen, tamoxifen, phenothiazines, or other vasodilators or antihypertensive agents such as guanethidine and derivatives within the last 12 months prior to Visit 2/Baseline.
    2. Any 5 alpha reductase medications (i.e., dutasteride, finasteride [Propecia®, etc.] or similar product[s]) within the last 12 months prior to Visit 2/Baseline.
    3. Retinoid therapy within the last 6 months prior to Visit 2/Baseline.
    4. Beta blockers, anabolic steroids, or corticosteroids (including intramuscular and intralesional injections) within 12 weeks of Visit 2/Baseline. Inhaled, intranasal, or ocular corticosteroids are allowed if use is stable (defined as doses and frequency unchanged for at least 4 weeks prior to Visit 2/Baseline.
    5. Drugs with antiandrogenic properties, such as flutamide, cimetidine, or ketoconazole within the last 6 months prior to Visit 2/Baseline; bicalutamide within 2 months and spironolactone within 1 month prior to Visit 2/Baseline. Gestagens with antiandrogen properties (e.g., cyproterone acetate, dienogest) are allowed if treatment is stable since the last 6 months prior to Visit 2/Baseline and if used as contraceptive.
    6. Minoxidil within the last 6 months prior to Visit 2/Baseline.
    7. Prostaglandins and derivates within the last 3 months prior to Visit 2/Baseline. Topical and ocular prostaglandins and its derivates are allowed.
    8. Biotin (>5 mg) within the last 4 weeks prior to Visit 2/Baseline.
    9. Previous radiation of the scalp and treatment with chemotherapy/systemic cytotoxic agents at any timepoint.
13. Participation in the evaluation of any investigational drugs within 30 days or 5 half lives (whichever is longer) prior to Visit 2/Baseline, calculated from the first day of the month following the last visit of the previous clinical trial.
14. History of drug and alcohol dependency.
15. In the opinion of the investigator the patient should not participate in the clinical trial, e.g., due to probable non compliance or inability to understand the clinical trial and give adequately informed consent.
16. Close affiliation with the investigator (e.g., a close relative) or persons working at the clinical trial centers or patient is an employee of sponsor.
17. Patient is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Target Area non vellus Hair Counts (TAHC) | From baseline to week 24
  This is the change in TAHC from Baseline to Week 24 (6 months). A descriptive analysis of the TAHC score at Baseline and Week 24 will be performed by treatment group (active, control and placebo). Also, a descriptive analysis of the change from Baseline to Week 24 (Week 24 - Baseline) will be performed by treatment group (active, control and placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Gómez-Sánchez, Study Director — Industrial Farmacéutica Cantabria, S.A.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carmina E, Azziz R, Bergfeld W, Escobar-Morreale HF, Futterweit W, Huddleston H, Lobo R, Olsen E. Female Pattern Hair Loss and Androgen Excess: A Report From the Multidisciplinary Androgen Excess and PCOS Committee. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2875-2891. doi: 10.1210/jc.2018-02548. PMID 30785992
- [Background] Russo PM, Fino E, Mancini C, Mazzetti M, Starace M, Piraccini BM. HrQoL in hair loss-affected patients with alopecia areata, androgenetic alopecia and telogen effluvium: the role of personality traits and psychosocial anxiety. J Eur Acad Dermatol Venereol. 2019 Mar;33(3):608-611. doi: 10.1111/jdv.15327. Epub 2018 Dec 2. PMID 30394586
- [Background] Olsen EA. Female pattern hair loss. J Am Acad Dermatol. 2001 Sep;45(3 Suppl):S70-80. doi: 10.1067/mjd.2001.117426. No abstract available. PMID 11511856
- [Background] Famenini S, Slaught C, Duan L, Goh C. Demographics of women with female pattern hair loss and the effectiveness of spironolactone therapy. J Am Acad Dermatol. 2015 Oct;73(4):705-6. doi: 10.1016/j.jaad.2015.06.063. No abstract available. PMID 26369846
- [Background] Starace M, Orlando G, Alessandrini A, Piraccini BM. Female Androgenetic Alopecia: An Update on Diagnosis and Management. Am J Clin Dermatol. 2020 Feb;21(1):69-84. doi: 10.1007/s40257-019-00479-x. PMID 31677111
- [Background] Redler S, Messenger AG, Betz RC. Genetics and other factors in the aetiology of female pattern hair loss. Exp Dermatol. 2017 Jun;26(6):510-517. doi: 10.1111/exd.13373. PMID 28453904
- [Background] Ramos PM, Brianezi G, Martins AC, da Silva MG, Marques ME, Miot HA. Apoptosis in follicles of individuals with female pattern hair loss is associated with perifollicular microinflammation. Int J Cosmet Sci. 2016 Dec;38(6):651-654. doi: 10.1111/ics.12341. Epub 2016 Jun 1. PMID 27163333
- [Background] Vano-Galvan S, Pirmez R, Hermosa-Gelbard A, Moreno-Arrones OM, Saceda-Corralo D, Rodrigues-Barata R, Jimenez-Cauhe J, Koh WL, Poa JE, Jerjen R, Trindade de Carvalho L, John JM, Salas-Callo CI, Vincenzi C, Yin L, Lo-Sicco K, Waskiel-Burnat A, Starace M, Zamorano JL, Jaen-Olasolo P, Piraccini BM, Rudnicka L, Shapiro J, Tosti A, Sinclair R, Bhoyrul B. Safety of low-dose oral minoxidil for hair loss: A multicenter study of 1404 patients. J Am Acad Dermatol. 2021 Jun;84(6):1644-1651. doi: 10.1016/j.jaad.2021.02.054. Epub 2021 Feb 24. PMID 33639244
- [Background] Shorter K, Farjo NP, Picksley SM, Randall VA. Human hair follicles contain two forms of ATP-sensitive potassium channels, only one of which is sensitive to minoxidil. FASEB J. 2008 Jun;22(6):1725-36. doi: 10.1096/fj.07-099424. Epub 2008 Feb 7. PMID 18258787
- [Background] Burton JL, Marshall A. Hypertrichosis due to minoxidil. Br J Dermatol. 1979 Nov;101(5):593-5. PMID 518830
- [Background] Zappacosta AR. Reversal of baldness in patient receiving minoxidil for hypertension. N Engl J Med. 1980 Dec 18;303(25):1480-1. doi: 10.1056/nejm198012183032516. No abstract available. PMID 7432414
- [Background] Jimenez-Cauhe J, Saceda-Corralo D, Rodrigues-Barata R, Moreno-Arrones OM, Ortega-Quijano D, Fernandez-Nieto D, Jaen-Olasolo P, Vano-Galvan S. Safety of low-dose oral minoxidil treatment for hair loss. A systematic review and pooled-analysis of individual patient data. Dermatol Ther. 2020 Nov;33(6):e14106. doi: 10.1111/dth.14106. Epub 2020 Sep 7. PMID 32757405